CLINICAL TRIAL: NCT06760845
Title: Research on Raman Spectroscopy Detection Technology in Kidney Disease Diagnosis
Brief Title: Raman Spectroscopy Diagnosis of Kidney Diseases
Status: Recruiting | Type: Observational
Sponsor: Zunsong Wang (Other)
Responsible Party: Sponsor-Investigator, Zunsong Wang, Dr, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: SERS-2024
Record Dates: First submitted 2024-12-12; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: IgA Nephropathy (IgAN); Membranous Nephropathy; Diabetic Nephropathy; Focal Segmental Glomerulosclerosis (FSGS)
MeSH Terms: conditions — Glomerulonephritis, IGA; Glomerulonephritis, Membranous; Diabetic Nephropathies; Glomerulosclerosis, Focal Segmental | interventions — Time-Lapse Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Imaging Time — Raman spectroscopy images of blood and urine

SUMMARY:
This research plan, from January 2021 to December 2024, aims to collect serum and morning urine from patients diagnosed with IgA nephropathy, idiopathic membranous nephropathy, diabetic nephropathy, and focal segmental glomerulosclerosis the Nephrology Department of Qianfoshan Hospital in Shandong Province, through renal biopsy. These samples will be scanned using a Raman spect to obtain Raman spectral data. The scattering peaks in the Raman spectra will be analyzed using Origin software for Gaussian curve fitting. The position of the peaks will used to query relevant literature to identify the corresponding chemical bonds and confirm the presence of compounds.

The intensity and area of the chemical substance peaks in the Raman will be calculated and used to plot calibration curves, thereby establishing a quantitative analysis equation. This equation will be used to accurately calculate the concentration of each analyte in serum and urine samples. Based on the average concentration data for each patient group, multivariate analysis methods, such as principal component analysis (PCA) and Mahalanis distance discriminant model, will be used to classify and predict the disease types.

The preliminary data for this study comes from the Nephrology Department ofianfoshan Hospital, where different types of glomerular diseases have been pathologically classified using tools such as light microscopy, electron microscopy, and immunoforescence microscopy. By combining Raman spectroscopy technology and statistical analysis, this study aims to establish a non-invasive and efficient diagnostic tool to assist in the of kidney diseases and predict treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Patients diagnosed with IgA nephropathy, idiopathic membranous nephrop, diabetic nephropathy, or focal segmental glomerulosclerosis confirmed by renal biopsy;
3. Patients who have not received hormone and/or immunosup therapy before the renal biopsy;

Exclusion Criteria:

1. Presence of factors causing secondary membranous nephropathy: such as autoimmune diseases (systemic lupus erythematosus),/infections (viral hepatitis), drugs or toxins, etc.;
2. Severe infection: clinical manifestations such as fever, cough and sputum, throat, abdominal pain, diarrhea, boils and other skin and soft tissue infections, with white blood cell count in blood routine exceeding the normal range (10×09/L);
3. Severe cardiovascular disease: including chronic heart failure of grade 3 or above and various arrhythmias;
4. Infect diseases: active phase of various types of hepatitis, AIDS, syphilis, etc.;
5. Evidence of tumor: already diagnosed with a certain tumor or manifestations, tumor markers, etc. indicating the possibility of a tumor;
6. Patients with incomplete data or missed diagnosis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Age 18 years or older;
  2. Patients diagnosed with IgA nephropathy, idiopathic membranous nephrop, diabetic nephropathy, or focal segmental glomerulosclerosis confirmed by renal biopsy;
  3. Patients who have not received hormone and/or immunosup therapy before the renal biopsy;
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Raman spectroscopy images of blood and urine | From the time of enrollment to the completion of blood and urine collection within 2 days
  The samples were scanned using a Raman spectrometer to obtain Raman spectral data. The scattering peaks in the Raman spectra were analyzed by fitting Gaussian curves using Origin software. The chemical bonds were identified and the presence of compounds was confirmed by referring to the literature based on the peak positions.
  The peak and area of the chemical substances in the Raman spectra were calculated and used to plot calibration curves, thereby establishing the quantitative analysis equation. This equation was used to calculate the concentrations of each analyte in the serum and urine.
  The average concentration data for each pathological patient group were used as the basis for multivariate analysis, such as principal component analysis (PCA) and Mahalanobis distance discriminant model, to classify and predict the types of diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Second Medical University. No.7166 Baotong West Street, Weifang, Shandong, 261053, China., Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Hematological and urinary biochemical indicators and Raman spectroscopic imaging

REFERENCES:
- [Background] Lima C, Muhamadali H, Goodacre R. The Role of Raman Spectroscopy Within Quantitative Metabolomics. Annu Rev Anal Chem (Palo Alto Calif). 2021 Jul 27;14(1):323-345. doi: 10.1146/annurev-anchem-091420-092323. PMID 33826853